CLINICAL TRIAL: NCT02600689
Title: Home-Based Pulmonary Rehab for Patients With Pulmonary Fibrosis
Acronym: EXPLORE-IPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Pulmonary Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, John D Lowman, PT, PhD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PFF-378875
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Pulmonary rehab; Exergame; Home-based
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical exercise training (Experimental): Combined aerobic and resistance exercise for 30 or more minutes at least 3 times per week for 12 weeks using the Wii Fit Plus
  Interventions: Behavioral: Physical exercise training
- Cognitive exercise training (Active Comparator): Cognitive, brain-training, video gaming ~30 minutes per session, 3 times per week for 12 weeks
  Interventions: Behavioral: Cognitive exercise training

INTERVENTIONS:
Behavioral: Physical exercise training
  Arms: Physical exercise training
Behavioral: Cognitive exercise training
  Arms: Cognitive exercise training

SUMMARY:
Outpatient (phase 2) pulmonary rehab is an important, but mostly underutilized intervention to improve physical function in patients with idiopathic pulmonary fibrosis (IPF). Of those individuals who complete phase 2 pulmonary rehab, only a small cohort continues with any type of maintenance exercise therapy (phase 3). This is largely due to personal factors, such as access to transportation, weather, scheduling difficulties, and cost.

Little is known about how to enhance physical activity among patients with IPF. In addition, no studies have investigated the long-term maintenance strategies of physical training in patients with IPF. Thus, the purpose of this study is to test the feasibility and effectiveness of a home-based, pulmonary rehab program for patients with IPF. A randomized, blinded, clinical trial (RCT) design with two arms -- Wii Fit Plus exergame program and cognitive video gaming, with no active whole body movement involved - will be used to investigate the benefits of a home-based exergame program on improving pulmonary-related function and symptoms in patients with IPF.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of IPF based on the criteria of the American Thoracic Society/European Respiratory Society 2011 guidelines;
* ≥ 40 years-of-age;
* ambulatory without the use of an assistive device;
* stable clinical condition (i.e., no pulmonary exacerbation for at least 6 weeks);
* no changes in medication for at least 4 weeks before enrollment;
* currently sedentary (i.e., exercise or participate in sports less than 3 times per week for 20 min in the past 6 months) and do not play any exergames;
* report dyspnea on exertion leading to a limitation in performing daily activities (i.e., Medical Research Council (MRC) dyspnea grade >1);
* able to read and follow exercise directions in English on the television screen;
* have permission from their treating physician to participate in moderate-intensity exercise;
* able to provide informed consent by understanding the nature of study participation.

Exclusion Criteria:

* contraindication for moderate-intensity exercise (e.g., unstable cardiac disease),
* severe musculoskeletal, vestibular, or neurological disorders limiting exercise performance, or inability to perform the 6-min walk test or 15-step test,
* requires > 6 lpm supplemental oxygen therapy via nasal cannula during exercise to maintain SpO2 >88%;
* MRC dyspnea grade 4 or 5; IPF patients with MRC dyspnea grade 4 or 5 have been reported to show little or no improvement, or deteriorated following pulmonary rehab;
* stage 2 hypertension,
* anemia (hemoglobin < 8 g/dL);
* collagen vascular disease;
* obstructive lung disease,
* non-parenchymal restrictive lung disease,
* occupational lung disease (pneumoconiosis, hypersensitivity pneumonitis),
* sarcoidosis,
* other idiopathic interstitial pneumonia;
* currently participating or have participated (in the past 30 days) in another clinical trial which can affect the outcomes of the proposed study; or
* planning to move out of Alabama within the next 6 months.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08; Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Functional performance | 12 weeks
  6-min walk distance (m)

SECONDARY OUTCOMES:
Exercise dyspnea | 12 weeks
  Dyspnea level (Borg CR10) after completing the 15-step test oximetry test
15-Step Test: Time | 12 weeks
  time (sec) to complete 15-step test
15-Step Test: Exercise desaturation | 12 weeks
  Level of desaturation (%) during 15-step test
15-Step Test: Recovery | 12 weeks
  Time to recovery to baseline oxygen saturation following 15-step test
Physical activity level | 12 weeks
  Time (min) spent per week in moderate-vigorous physical activity (assessed via an accelerometer)
Health-related quality of life | 12 weeks
  St George's Respiratory Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hon K Yuen, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Yuen HK, Lowman JD, Oster RA, de Andrade JA. Home-Based Pulmonary Rehabilitation for Patients With Idiopathic Pulmonary Fibrosis: A PILOT STUDY. J Cardiopulm Rehabil Prev. 2019 Jul;39(4):281-284. doi: 10.1097/HCR.0000000000000418. PMID 31241519